CLINICAL TRIAL: NCT07214610
Title: Carolina Breast Cancer Study: Integrating Biological, Clinical, and Behavioral Factors to Improve Breast Cancer Outcomes in the Carolina Breast Cancer Study, Phase 4
Brief Title: Integrating Biological, Clinical, and Behavioral Factors to Improve Breast Cancer Outcomes - Carolina Breast Cancer Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other); Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-0956
Record Dates: First submitted 2025-10-08; First posted 2025-10-09 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: subtypes of breast cancer; genetic factors; racial disparities; African American (AA); American Indian/Alaska Native (AIAN); tumor biology; treatment adherence; patient engagement
MeSH Terms: conditions — Breast Neoplasms; Treatment Adherence and Compliance; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Newly diagnosed with breast cancer (Experimental): Participants with newly diagnosed with breast cancer live in 59 North Carolina counties.
  Interventions: Behavioral: Structured behavioral intervention

INTERVENTIONS:
Behavioral: Structured behavioral intervention — All participants will be prospectively assigned to a structured behavioral intervention embedded within the research process. The goal of the intervention is to improve communication with healthcare providers and enhance self-advocacy during breast cancer care. Components include reflective behavioral self-assessments, symptom reporting tools, regular interaction with nurses and lay health educators, access to webinars and newsletters, patient-centered educational materials, and the return of study results to participants through a report-back process. The behavioral engagement components are standardized and delivered over the first 12 months post-enrollment.
  Other Names: Structured behavioral intervention embedded within the research process

SUMMARY:
Phase 4 of the Carolina Breast Cancer Study (CBCS4) builds on prior phases that examined molecular and epidemiologic differences in breast cancer types and outcomes. Previous findings showed that certain breast cancer subtypes and genetic factors are linked to higher risks. While prior research uncovered subtype-specific risks and relevant genetic loci, persistent disparities especially among African American (AA) and American Indian/Alaska Native (AIAN) women suggest that tumor biology alone does not fully explain outcome differences. Other important factors, like access to healthcare, treatment adherence, patient engagement must also be evaluated.

In addition to collecting biological and clinical data, participants will receive a structured behavioral intervention designed to improve communication with providers and self-advocacy during cancer care. This phase includes a structured behavioral intervention designed to improve health communication and self-advocacy, both of which are hypothesized to improve health outcomes. All participants are prospectively assigned to this single-arm intervention, which includes educational resources, symptom reporting tools, reflective self-assessments, and regular engagement with trained study staff over a defined timeline.

This study assesses whether structured research participation can positively influence patient behavior and ultimately reduce disparities in breast cancer care.

This study also aims to better understand etiology and prognosis of breast cancer, including subtypes such as Luminal A and B, Basal-like, and Human Epidermal Growth Factor Receptor 2 positive (HER2+) / estrogen receptor negative (ER-) and to address disparities driven by both biology and systemic barriers.

DETAILED DESCRIPTION:
Study Population will be 3300 participants with invasive breast cancer among women aged 20-74 in 59 North Carolina counties between will be enrolled. Approximately 1,500 Black women (750 aged <50 and 750 aged ≥50) and 1,750 non-Black women, including approximately 200 who self-identify as American Indian/Alaska Native (875 <50, 875 ≥50) will be included.

Participants will complete a structured, in-person baseline interview covering breast cancer risk factors, quality of life, comorbidities, initial treatment, follow-up surveys will assess changes in self advocacy. Blood and/or saliva samples will be collected. Participants will provide consent for medical record abstraction and retrieval of tumor blocks.

ELIGIBILITY:
Inclusion Criteria:

* women with invasive breast cancer
* live in 59 counties in North Carolina

Exclusion Criteria:

* women with ductal carcinoma in situ (DCIS)
* live outside of 59 counties of North Carolina

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3300 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2044-12-31 (Estimated); Study Completion 2044-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Communication Self-Efficacy Score | Baseline, 19 months, every 12-24 months up to 15 years
  Patient communication self-efficacy will be measured using the Patient's Communication Perceived Self-Efficacy Scale (PCSS), a validated patient-reported instrument comprising 16 items with a three-factor structure: Provide and Collect Information, Express Concerns and Doubts, and Verify Information. The scale assesses patients' confidence in their ability to communicate effectively with healthcare providers about health concerns, ask questions, express uncertainties, and confirm their understanding. Items are rated on a 5-point Likert scale (1 = not at all confident to 5 = very confident), with total scores ranging from 16 to 80. Higher scores indicate greater perceived communication self-efficacy.

SECONDARY OUTCOMES:
Tumor Recurrence Events | 9 months, 19 months, every 12-24 months up to 15 years
  Tumor recurrence will be identified via electronic medical records based on clinical documentation of local, regional, or distant recurrence of the primary cancer. The date and location of recurrence will be recorded using standardized clinical criteria.
Incidence of Second Primary Tumors | 9 months, 19 months, every 12-24 months up to 15 years
  Second primary tumors will be identified through electronic medical records and pathology reports. Criteria for classification as a second primary cancer and date of diagnosis will follow standard oncology definitions, distinct from recurrence of the original tumor.
Breast Cancer-Specific and All-Cause Mortality | 8 years and 15 years
  Mortality data, including breast cancer-specific and all-cause mortality, will be collected from electronic medical records and/or linked national death registries. Information will include vital status, cause of death, and date of death.
  Time Frame:
Quality of life measured using the Functional Assessment of Cancer Therapy - Breast (FACT-B) | 9 months, 19 months, every 12-24 months up to 15 years
  Quality of life will be assessed using the Breast (FACT-B) which is a validated, patient-reported outcome measure designed to assess quality of life in individuals with breast cancer. It combines the general FACT-G (Functional Assessment of Cancer Therapy - General) questionnaire with a breast cancer-specific subscale. The tool evaluates five domains: physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns specific to breast cancer. The FACT-B consists of 37 items, combining the 27-item FACT-G (general quality of life) and a 10-item Breast Cancer Subscale (BCS). Each item is rated on a 5-point Likert scale from 0 (not at all) to 4 (very much). Higher scores indicate better quality of life.
Quality of life measured using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | 9 months, 19 months, every 12-24 months up to 15 years
  Quality of life will be assessed using the EORTC QLQ-C30 is a cancer-specific instrument with 30 questions which incorporates 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 9 symptom scales (fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties); and a global health and quality-of-life scale. Most questions used 4 point scale (1 'Not at all' to 4 'Very much'); 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). The scores of these scales were averaged from the scores of the component items, transformed and analyzed on a 0 - 100 scale. A higher score=better level of functioning or greater degree of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials